CLINICAL TRIAL: NCT02971722
Title: Randomized,Double-blind,Placebo-controlled,Dose-escalating Phase I,Healthy Subjects Study of JY09,a Recombinant GLP-1 Receptor Agonist
Brief Title: a Study of JY09 in Chinese Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Dongfang Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFBT-JY09-1
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: GLP-1 receptor agonist

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 0.3mg JY09(cohort 1) (Experimental): 0.3mg JY09 administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: JY09
- 1.5mg JY09(cohort 1) (Experimental): 1.5mg JY09 administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: JY09
- 6.0mg JY09(cohort 1) (Experimental): 6.0mg JY09 administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: JY09
- Placebo(cohort 1) (Placebo Comparator): Placebo administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: Placebo
- 0.7mg JY09(cohort2) (Experimental): 0.7mg JY09 administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: JY09
- 3.0mg JY09(cohort2) (Experimental): 3.0mg JY09 administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: JY09
- 12.0mg JY09(cohort2) (Experimental): 12.0mg JY09 administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: JY09
- Placebo(cohort 2) (Placebo Comparator): Placebo administered once subcutaneous injection to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JY09 — 2mg/1ml/bottle
  Arms: 0.3mg JY09(cohort 1); 0.7mg JY09(cohort2); 1.5mg JY09(cohort 1); 12.0mg JY09(cohort2); 3.0mg JY09(cohort2); 6.0mg JY09(cohort 1)
Drug: Placebo — 1ml/bottle
  Arms: Placebo(cohort 1); Placebo(cohort 2)

SUMMARY:
JY09，is a recombinant glucagon-like peptide-1 (GLP-1) receptor agonist,constructed with Exendin-4 and human Immunoglobulin G2 (IgG2) Fc fragment.Preclinical studies show that JY09 exhibit the expected GLP-1-mediated pharmacological effects on insulin secretion,glucose covering and islet cell recovering,as well as good tolerance and safety.JY09 has been approved by China food and drug administration(CFDA) to enter the clinical research stage(Grant number 2016L04254).This study is designed to assess the safety,tolerability,pharmacokinetics,pharmacodynamics and potential immunogenicity of JY09 in healthy Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects.
* Male's mass is equal or greater than 50 kg, female's mass is equal or greater than 45 kg,have a body mass index (BMI) between 18 and 28 kilograms per square meter (kg/m^2), inclusive.
* The subjects sign informed consent form voluntarily.
* The subjects agree to use instruments of contraception from the time of the first dose until 6 months after the last dose of investigational drug, avoid pregnancy make yourself or your mate.
* Participants will be able to keep good communication with investigator and comply with the requirements of the clinical trials

Exclusion Criteria:

* Smokers,quitting time less than 3 months , or can't quit smoking during the trial.
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing,or being treated for a direct lower gastrointestinal or using steroids.
* Participation in any clinical investigation within 3 months prior to dosing
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing
* Significant illness within 2 weeks prior to dosing,and investigator judge doesn't fit to participate in this trial.
* A history of clinical significance of abnormal ECG or family history of long QT syndrome (grandparents, parents and siblings)
* Have a family history of diabetes (grandparents, parents and siblings).
* Have a history of acute or chronic bronchial spasms(including after treatment or no treatment of asthma and chronic obstructive pulmonary disease )
* Have a history of drug allergy or atopic disease allergy(asthma, urticaria, eczema, dermatitis),or allergy history of trail drugs or similar drugs.
* Have gastrointestinal diseases,such as history of liver disease, gastrointestinal disease,gastrointestinal surgery (appendix removed except) or chronic pancreatitis, or history of idiopathic acute pancreatitis that,in the opinion of the investigator,is clinical significant.
* Have personal or family history of medullary thyroid cancer (MTC) or a hereditary disease that induce MTC .
* Have a history of immunodeficiency disease,including human immunodeficiency virus (HIV) antibody positive.
* Have a history of needlesickness that,in the opinion of the investigator,is clinical significant.
* Have an unknown cause of infection.
* In screening,any abnormal results of physical examination, vital signs,electrocardiogram (ECG) and clinical laboratory that,in the opinion of the investigator,is clinical significant.
* Hepatitis b surface antigen or hepatitis c antibody positive, or treponema pallidum antibody positive.
* Abuse of drug or alcohol within 12 months before first dosing,or in screening found evidence of abuse in laboratory tests.
* People who are pregnant, nursing mothers, or in the near future plan to be pregnant,or show pregnancy test positive before into group.
* In screening,lying position (after 3 minutes rest) systolic blood pressure outside the range 90 ~ 140 MMHG, or diastolic blood pressure outside the range 50-90 MMHG, or pulse (HR) outside the range 40 ~ 100 bpm, boundary value into the group.
* Have chang of weight > 3 kg within 3 months by self-report.
* Subjects who, in the opinion of the investigator, are in any way unsuitable to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) | Baseline through day29 of period
  Area Under the Concentration Versus Time Curve (AUC) of JY09

SECONDARY OUTCOMES:
immunogenicity | Baseline through day29 of period
  A measure of the body's immune response to JY09
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | baseline to 3 months(cohort1 and cohort 2)
  Weight loss of subject is greater than 3 kg will be recorded as adverse events in a month
Pharmacodynamics (PD） | Baseline through day29 of period
  Area Under the Concentration Versus Time Curve (AUC) of Glucose

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorkildsen C, Neve S, Larsen BD, Meier E, Petersen JS. Glucagon-like peptide 1 receptor agonist ZP10A increases insulin mRNA expression and prevents diabetic progression in db/db mice. J Pharmacol Exp Ther. 2003 Nov;307(2):490-6. doi: 10.1124/jpet.103.051987. Epub 2003 Sep 15. PMID 12975499
- [Background] Bradley DP, Kulstad R, Schoeller DA. Exenatide and weight loss. Nutrition. 2010 Mar;26(3):243-9. doi: 10.1016/j.nut.2009.07.008. PMID 20152707